CLINICAL TRIAL: NCT06492161
Title: Evaluation of an Application Allowing Physical Activity to Get Information on Their Physical Activity in the First Days Following Thoracic Surgery
Brief Title: Physical Activity Measure Application
Acronym: MARCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020_0140
Record Dates: First submitted 2024-06-24; First posted 2024-07-09 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Physical Inactivity; Post-Surgical Complication
Keywords: ActiGraph GT3X; Physical activity; Thoracic surgery; ACTIM application
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT3X ActiGraph's activity monitor (Experimental): Patients who have undergone thoracic surgery wearing an ActiGraph GT3X-BT device that measures and records physical movement associated with daily activity.
  Interventions: Device: Physical activity measure

INTERVENTIONS:
Device: Physical activity measure — After surgery, patients patients will be fitted with GT3X ActiGraph's activity monitor to capture and record continuous physical activity.

SUMMARY:
Although there is a strong physiological rationale for the benefit of post-operative mobilization, the evidence supporting these effects in surgical cohorts is conflicting, and there is a lack of research to guide the clinical implementation of early mobilization protocols. There is also a need to better evaluate the physical activity performed by physical activity tients outside the supervised mobilization protocol, to better understand its potential benefits on post-operative recovery. In adition, the objective measurement of physical activity has several advantages over declarative measures.

DETAILED DESCRIPTION:
Prolonged immobilization after surgery is known to have detrimental effects. Although postoperative recommendations favor early mobilization, the lack of quantification of physical activity poses a problem for the implementation of early mobilization protocols..

An application named "ACTIM" has been developed with the aim of automating the personalized assessment of postoperative physical activity. The healthcare team (nurses or physiotherapists…), will share the information with the patient and will complete the assessment using personalized physical activity objectives for the day.

The purpose of this study is to assess this application in real-life settings to provide patients with information on their physical activity after lung resection by thoracoscopy or robotic surgery. This assessment will serve as a reference for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Scheduled for thoracoscopic or robotic lung resection
* Agreeing to wear an ActiGraph GT3X accelerometer from 4 days post-surgery
* Having signed a consent form
* Affiliated with a health insurance

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient unable to move independently (paraplegic, etc.)
* Patient deprived of liberty or under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Assess the agreement between ACTIM application and Actilife Softawre for the sitting-lying position | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of time spent sitting/lying-down
Assess the agreement between ACTIM application and Actilife Softawre for sitting-standing transition | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of number of sit-to-stand transitions
Assess the agreement between ACTIM application and Actilife Softawre for step count | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of number of number of steps
Assess the agreement between ACTIM application and Actilife Softawre for walking pace | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of number of walking cadence

SECONDARY OUTCOMES:
Measuring changes in physical activity with ACTIM application from postoperative Day 1 up to Day 4 | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of time spent sitting/lying-down using ACTIM application
Measuring changes in physical activity with ACTIM application from postoperative Day 1 up to Day 4 | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of number of sitting-standing transition using ACTIM application.
Measuring changes in physical activity with ACTIM application from postoperative Day 1 up to Day 4 | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of step count using ACTIM application.
Measuring changes in physical activity with ACTIM application from postoperative Day 1 up to Day 4 | up to 4 days
  Measure, from postoperative Day 1 up to Day 4 of walking pace using ACTIM application.
Measuring changes in physical activity with Actilife Softawre from postoperative Day 1 up to Day 4 | up to 4 days
  Measure of indicators of physical activity volume :
  Number of counts/day (Sum of counts (vertical axis) accumulated over the day) Number of steps/day (Sum of steps accumulated over the day)
Measuring changes in physical activity with Actilife Softawre from postoperative Day 1 up to Day 4 of physical activity intensity | up to 4 days
  Measure of indicators of physical activity intensity :
  Average number of counts/minute, Average walking pace (Average number of steps/minute).
Measuring changes in physical activity with Actilife Softawre from postoperative Day 1 up to Day 4 of duration | up to 4 days
  Measure of Indicators of duration :
  Sedentary time (Total minutes/day < 100 counts/minute), Light-intensity physical activity (Total minutes/day between 100 and 1,951 counts/minute), Moderate-intensity physical activity (Total minutes/day between 1,952 and 5,724 counts/minute), High-intensity physical activity (Total minutes/day ≥ 5,725 counts/minute), Moderate/high-intensity physical activity (Total minutes/day ≥ 1,952 counts/minute).
Measuring changes in physical activity with Actilife Softawre from postoperative Day 1 up to Day 4 of duration of walking at each intensity | up to 4 days
  Measure of indicators of duration of walking at each intensity :
  Occasional movement (Number of minutes with 1 to 19 steps/minute), Sporadic movement (Number of minutes with 20 to 39 steps/minute), Intentional walking (Number of minutes with 40 to 59 steps/minute), Slow walking (Number of minutes with 60 to 79 steps/minute), Moderate walking (Number of minutes with 80 to 99 steps/minute), Brisk walking (Number of minutes with 100 to 119 steps/minute), Fast walking (Number of minutes with ≥ 120 steps/minute),
Measuring changes in physical activity with Actilife Softawre from postoperative Day 1 up to Day 4 of energy expenditure | up to 4 days
  Measure of indicators of energy expenditure : physical activity-related energy expenditure estimated by a prediction equation
Measuring changes in physical activity with Actilife Softawre from postoperative Day 1 up to Day 4 of moderate to high-intensity physical activity | up to 4 days
  Measure of indicators of moderate to high-intensity physical activity :
  Number of sessions/day (Number of sessions (≥ 1 min) ≥ 1,952 counts/minute), Average session duration (Average session duration ≥ 1,952 counts/minute), Number of sessions ≥ 10 min (Number of sessions (≥ 10 min) ≥ 1,952 counts/minute), Total duration in sessions ≥ 10 min (Total duration of physical activity in sessions ≥ 10 min).
Measuring changes in physical activity with Actilife Softawre from postoperative Day 1 up to Day 4 of sedentary | up to 4 days
  Measure of indicators of sedentary :
  Number of sessions/day (Session number (≥ 1 min) < 100 counts/minute), Average session duration (Average duration of sessions < 100 counts/minute), Number of sessions ≥ 10 min (Session number (≥ 10 min) < 100 counts/minute), Total duration in sessions ≥ 10 min (Total duration of sedentary behavior in sessions ≥ 10 min),
Assess of the practical feasibility and level of satisfaction of the medical team regarding the personalized assessment obtained through ACTIM application | up to 4 days
  The level of satisfaction/feasibility with the ACTIM application will be assessed using a satisfaction scale from 0 to 10 (0: Not satisfactory and 10: Very satisfactory) when the device will be remove.
Record patients' interest in the format and information contained in the personalized report | up to 4 days
  Using an interest scale from 0 to 10 (0: Not interesting to 10: Very interesting). The format in which this information is made available will be evaluated using a satisfaction scale (0: Not satisfactory to 10: Very satisfactory) when the device will be remove.
Record postoperative complications | up to 4 days
  Postoperative complications will be recorded using the 'Morbidity and Mortality after Thoracic Surgery' classification from hospital discharge up to 1 month post surgery
Assess patient acceptability of wearing the ActiGraph GT3X | up to 4 days
  Patients' acceptability of wearing the ActiGraph GT3X will be assessed when the equipment is removed, using a simple numerical scale ranging from 0 : unbearable to wear to 10 : no discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Julien FESSLER, MD, Principal Investigator — Foch Hospital
Locations (1):
- Foch Hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Background] Ljungqvist O. ERAS--enhanced recovery after surgery: moving evidence-based perioperative care to practice. JPEN J Parenter Enteral Nutr. 2014 Jul;38(5):559-66. doi: 10.1177/0148607114523451. Epub 2014 Feb 24. PMID 24567343
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Chomistek AK, Yuan C, Matthews CE, Troiano RP, Bowles HR, Rood J, Barnett JB, Willett WC, Rimm EB, Bassett DR Jr. Physical Activity Assessment with the ActiGraph GT3X and Doubly Labeled Water. Med Sci Sports Exerc. 2017 Sep;49(9):1935-1944. doi: 10.1249/MSS.0000000000001299. PMID 28419028
- [Background] Daskivich TJ, Houman J, Lopez M, Luu M, Fleshner P, Zaghiyan K, Cunneen S, Burch M, Walsh C, Paiement G, Kremen T, Soukiasian H, Spitzer A, Jackson T, Kim HL, Li A, Spiegel B. Association of Wearable Activity Monitors With Assessment of Daily Ambulation and Length of Stay Among Patients Undergoing Major Surgery. JAMA Netw Open. 2019 Feb 1;2(2):e187673. doi: 10.1001/jamanetworkopen.2018.7673. PMID 30707226
- [Background] Seely AJ, Ivanovic J, Threader J, Al-Hussaini A, Al-Shehab D, Ramsay T, Gilbert S, Maziak DE, Shamji FM, Sundaresan RS. Systematic classification of morbidity and mortality after thoracic surgery. Ann Thorac Surg. 2010 Sep;90(3):936-42; discussion 942. doi: 10.1016/j.athoracsur.2010.05.014. PMID 20732521